CLINICAL TRIAL: NCT06409416
Title: Identification of Molecular Mechanisms Which Drive Tumor Cell Plasticity and Aggressiveness in Human Non-small Cell Lung Cancer
Brief Title: Tumor Cell Plasticity and Aggressiveness in Human Non-small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Fabrizio Bianchi, Head, cancer Biomarkers Unit, Casa Sollievo della Sofferenza IRCCS
Other Study IDs: RF-2021-12372433
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Lung Neoplasms; Progression
MeSH Terms: conditions — Lung Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of diagnostic biomarkers — The investigators will analyze TCP-biomarkers diagnostic by IHC, qRT-PCR and next-generation sequencing, in tumor and plasma samples of lung cancer patients.

SUMMARY:
Tumor cell plasticity (TCP) is a conubium of processes which lead to re-activation of developmental programs correlating with epithelial-to-mesenchymal transition, and ultimately leading to acquisition of stem cell properties and transdifferentiation potential. Little is known about the molecular mechanisms governing TCP in lung adenocarcinoma (LUAD), i.e. the most frequent lung cancer subtype. The investigators recently identified prognostic 7-miRNAs/10-mRNAs signatures which accurately identified aggressive LUAD among patients with early-stage disease (Stage I). Furthermore, the investigators showed that such tumors show TCP features i.e. mesenchymal and stem-cell traits, high-metastatic potential. Here, the investigators aim to explore by RNAseq and by immunophenotyping at a single-cell level (scRNAseq/AbSeq), the molecular features of aggressive LUAD to unveil the mechanisms triggering TCP. The investigators predict thier results will be relevant for the development of more effective therapeutic protocols for management of aggressive LUAD.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with lung adenocarcinoma
* treatment naive
* undergoing primary surgery

Exclusion Criteria:

* patients with a previous history of cancer
* previously treated by chemio/immuno/radio-therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing surgery for confirmed diagnosis of lung adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
TCP-biomarkers screening in a prospective cohort of lung cancer patients | 36 months
  The investigators will: i) deconvolute the tumor epithelial cell heterogeneity of lung adenocarcinoma (LUAD) by coupling immunophenotype screening and single-cell RNAseq profiling of human LUAD samples; ii) identify subsets of LUAD cells with "active" tumor cell plasticity (TCP) using both our miRNA/RNA prognostic signatures, the C1-LUAD geneset (N=330), and previously identified signatures of lung cells high-cell plasticity (HCP) state; iii) explore the molecular features of TCP cell subsets by gene-network rewiring, pathway reconstruction analysis, and functional validation experiments of molecular "HUBs" controlling TCP pathways. Biomarkers of TCP will be also prioritized among TCP-hallmark genes and validated by immunohistochemistry (IHC/FACS) in human LUAD.